CLINICAL TRIAL: NCT00972972
Title: Effect of Bilberry (European Blueberries) and Grape Polyphenols on Cognition and Blood Parameters in Normal, Aged Men With Subjective Memory Decline
Brief Title: Effect of Bilberry (European Blueberries) and Grape Polyphenols on Cognition and Blood Parameters
Acronym: BLUEBERRY
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Ulleval University Hospital, Ulleval University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 699
Record Dates: First submitted 2009-09-03; First posted 2009-09-09 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Memory; Gene Expression
Keywords: fruit polyphenols; phytochemicals; neurocognition; neuropsychology; psychopharmacology; gene expression; biochemistry
MeSH Terms: interventions — Vaccinium myrtillus extract; Polyphenols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dietary supplement (Active Comparator): Extracts of bilberry (European blueberries) and red grape juice (Merlot grapes; Vitis Vinifera L.)
  Interventions: Dietary Supplement: bilberry (European blueberries) and red grape juice
- placebo dietary supplement (Placebo Comparator): Placebo juice extracts
  Interventions: Dietary Supplement: placebo juice

INTERVENTIONS:
Dietary Supplement: bilberry (European blueberries) and red grape juice — Intervention juice: 50/50 combination of 300 ml bilberry (European blueberries) and red grape juice (Merlot grapes; Vitis Vinifera L.) per day for 9 weeks
  Other Names: Bilberry; European blueberries; polyphenols
  Arms: dietary supplement
Dietary Supplement: placebo juice — Placebo juice: 300 ml, similar to the intervention juice as to taste, energy, salt, and carbohydrates
  Arms: placebo dietary supplement

SUMMARY:
The purpose of this study is to determine whether dietary intervention with blueberry and grape juice extracts in elderly men with subjective memory problems would raise performance on neuropsychological memory tests and change biomarker of muscle damage and whole blood gene expression profiles.

DETAILED DESCRIPTION:
A number of studies have shown that increased dietary intake of fruits and vegetable extracts high in antioxidants (e.g., blueberries, strawberries and spinach) can retard and even reverse age-related decline in brain function and in cognitive and motor performance in rats. This is the first placebo-controlled human study to evaluate the effect of dietary intake of fruit polyphenols on neuropsychological test scores and whole blood gene regulation

Sixty-two non-demented, non-depressed men (age 67-77 years) with subjective memory decline, were randomly assigned to a blueberry/grape juice- and placebo-group in a 9 week double blind intervention study. Pre- and post treatment assessment were measured with a computerised neuropsychological test battery (CANTAB), including tests for motor speed, visual reaction time, and spatial memory. Dietary habits were registered before intervention and several clinical biomarkers were measured in plasma/serum before and after the intervention. Pre- and post intervention-samples for measurement of gene regulation were also collected

ELIGIBILITY:
Inclusion Criteria:

* men
* age 67-77 years
* gradual subjective memory decline
* response to advertisement

Exclusion Criteria:

* head trauma with loss of consciousness and lasting symptoms
* brain stroke within last 3 years
* dementia, clinically diagnosed
* signs of brain-degenerative disease
* Mini Mental Status Examination score less than 26
* depression (MADRS; Montgomery Asberg Depression Rating Scale score above 20)
* ongoing treatment for cancer (cytostatica)/diabetes
* reported or observed serious mental illness
* reported or observed use of narcotics (any, present or past)
* reported or observed abuse of alcohol
* visual, auditory, or motor handicaps of relevance for performance

Ages: 67 Years to 77 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-12; Primary Completion 2007-07 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
neuropsychological test scores and whole blood gene regulation | December 2006 - july 2007
whole blood gene regulation; parameters in blood | 2006 and 2007
neuropsychological test scores; whole blood gene regulation; parameters in blood | 2006 and 2007

SECONDARY OUTCOMES:
gene expression of stress, repair and maintenance processes measured by whole genome microarray analysis in blood | 2007 and 2009

CONTACTS AND LOCATIONS:
Overall Officials: KJELL - FLEKKOY, DR. PHILOS., Principal Investigator — ULLEVAAL UNIVERSITY HOSPITAL; UNIVERSITY OF OSLO; RUNE - BLOMHOFF, DR. MED., Principal Investigator — University of Oslo
Locations (1):
- Ulleval University Hospital HF, Oslo, Norway

REFERENCES:
- [Derived] Bohn SK, Myhrstad MCW, Thoresen M, Erlund I, Vasstrand AK, Marciuch A, Carlsen MH, Bastani NE, Engedal K, Flekkoy KM, Blomhoff R. Bilberry/red grape juice decreases plasma biomarkers of inflammation and tissue damage in aged men with subjective memory impairment -a randomized clinical trial. BMC Nutr. 2021 Nov 22;7(1):75. doi: 10.1186/s40795-021-00482-8. PMID 34802467